CLINICAL TRIAL: NCT06609044
Title: Social and Psychological Long-term Impact of NMDA Receptor Encephalitis
Brief Title: Long-term Impact of NMDAR Encephalitis
Acronym: SAPIENCE2
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0793; 2024-A01958-39 (Other: ID-RCB)
Record Dates: First submitted 2024-09-06; First posted 2024-09-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Autoimmune Encephalitis
Keywords: NMDAR encephalitis; psychosocial impact
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anti-NMDAR encephalitis patients.: Patients over 18 years old with NMDAR encephalitis.

SUMMARY:
NMDA receptor antibody encephalitis is a rare autoimmune neurological disease of the central nervous system with an estimated incidence of 1.5 people per million per year. Patients with anti-NMDAR encephalitis experience an acute phase of the disease characterized by psychosis, memory loss, seizures, autonomic nervous system instability, or coma. Since the discovery of this disease 14 years ago by Prof. Dalmau, the clinical presentation of the acute phase has been well characterized, while the psychosocial impact of the disease remains largely unexplored.

Currently, there are few cohort studies of patients that have identified persistent cognitive impairment as a factor impacting remission after the acute phase. Given the scarcity of information concerning the post-acute phase, it is therefore essential to determine the long-term social and psychological outcomes and their daily effects on the social and functional life of this severe disease. This is especially important as the patients are young, with a median age of 21 years, and may face lasting limitations potentially detrimental to their success in professional, educational, or social environments.

DETAILED DESCRIPTION:
This study will help improve the management of patients with anti-NMDAR encephalitis :

* By providing the first assessment of long-term cognitive, psychological and social consequences
* By characterizing the patient's journey through the disease
* By developing a standardized neuropsychological assessment which will improve the assessment of the patient in the post-acute phase As well as improving patient care in the long term through the drafting of specific medical recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NMDAR encephalitis
* Age ≥ 18 years old
* Patient affiliated to a social security system
* No opposition from the patient

Exclusion Criteria:

* Patients whithout NMDAR encephalitis
* Age < 18 years old
* Patient under guardianship or curatorship
* Patient with neurological disorders pre-existing encephalitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anti-NMDA encephalitis aged over 18 years old and followed in Lyon.
  We plan to include 30 patients.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Psychosocial questionnaires of patients with anti-NMDAR encephalitis after the acute phase of the disease. | 50 MINUTES
  Neuropsychological Questionnaires :
  * RAVLT questionnaire (no score)
  * EMPAN questionnaire (no score)
Analysis of cognitive assessments of patients with anti-NMDAR encephalitis after the acute phase of the disease. | 40 MINUTES
  Score of PROMs questionnaires :
  * FSS (score : /63)
  * HADS (score : /42)
  * EQ5D5L (score : /100)
  * BDI-II (no score )
  * MMQ (no score)
  * PSQI (no score)
Patient's experience of the disease | 1 Year
  Score of Clinical questionnaire about patient's experience of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme HONNORAT, MD, Principal Investigator — Centre de référence des syndromes neurologies paranéoplasiques et encéphalites auto-immunes - Hôpital neurologiques Pierre WERTHEIMER - Groupement hospitalier Est - Hospices civiles de Lyon
Locations (1):
- Centre de référence des syndromes neurologies paranéoplasiques et encéphalites auto-immunes - Hôpital neurologiques Pierre WERTHEIMER, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boeken OJ, Heine J, Duda-Sikula M, Patricio V, Picard G, Buttard C, Benaiteau M, Mendes A, Howard F, Easton A, Kurpas D, Honnorat J, Dalmau J, Finke C. Assessment of long-term psychosocial outcomes in N-methyl-D-aspartate receptor encephalitis - the SAPIENCE study protocol. BMC Neurol. 2024 Sep 6;24(1):322. doi: 10.1186/s12883-024-03842-6. PMID 39242986